Title: The assessment of fatigue and quality of life in patients with bone tumor, undergoing chemotherapy treatment and possible predictive factors.

Code: Fatigue-ONCO

**Sources of financing**: this study is a spontaneous non-profit study

**Conflict of interest:** No conflict of interest on the part of the principal investigator, nor of

the Collaborators

Principal Investigator: Dr.ssa Paola Coluccino, SSD Chemioterapia

Firma del PI

**Promotor:** Istituto Ortopedico Rizzoli – SSD Chemioterapia

# Co investigator:

Mattia Morri, Physiotherapist, Physical and Rehabilitative medicine

Rita Boschi, Nurse, Chemotherapy ward

Eugenio Brruku, Nurse, Chemotherapy ward

Erika Romagnoli, Nurse, Chemotherapy ward

Riccardo Boccomino, Nurse, Chemotherapy ward

### Acronyms used in the text

**BFI:** Brief Fatigue Inventory

**EORTC QLQ C-30** 

**TESS:** Toronto Extremity Salvage Score

Ver.1.0 del 30/04/2019 1/11

**BMI:** Body mass index

**NRS**: Numering Rate Scale

**CRF:** Case Report Form

Introduction

Fatigue syndrome is defined as an altered physical, emotional and / or cognitive

feeling of tiredness that is not proportional to the activities performed by the

subject and interferes with the activity of daily life (NCCN, 2018, Bower, 2014). It is a

clinical condition, linked to the oncological pathology, extremely widespread and in

patients undergoing chemotherapy and / or radiotherapy it is common in 80% of patients

(NCCN, 2018; Bower, 2014; Arajuo, 2017).

At the same time this symptomatology is identified as under-estimated and under-treated.

Hubbard et al (2014), in accordance with the guidelines, suggest the need to introduce

assessment of fatigue as a screening element for normal clinical practice. Interventions

aimed at increasing physical activity, psychosocial and pharmacological support can

benefit patients even if a standard treatment model has not been described to date

(Bower, 2014). One of the difficulties highlighted in the literature is the correct identification

of this syndrome. Scott et al (2011) stress the need for systematic studies in cancer

populations with different types of cancer and at different stages of the disease using

patient-oriented fatigue assessment tools. The Brief Fatigue Inventory (BFI) is one of the

scales used precisely in the evaluation of this syndrome and has proved to be a reliable

and easy to use tool, also validated in Italian (Mendoza et al 1999, Catania et al. 2013).

Several authors have also shown that reduced physical activity and a worse quality of life

are associated with fatigue (Witt et al 2002; Stark et al 2012, Warner et al 2008),

particularly in young patients (Poort et al 2017).

In the area of bone tumors, the available data on fatigue syndrome are extremely poor and

only two studies have emerged from the literature search. The study by Granada-Cameron

et al (2011) describes the experience of 11 new sarcoma patients undergoing

chemotherapy treatment. Fatigue had been described as the prevalent symptom and was

related to a worse quality of life.

Serveas et al (2003) observing patients two years after the conclusion of treatment for

bone cancer found that in 28% of cases fatigue is a severe problem for patients.

Objective

The aim of the present study is to evaluate and describe the evolution over time of the

fatigue and the quality of life of patients with bone tumor during the chemotherapy

treatment and in the first phase of follow-up and to identify possible prognostic factors.

Such knowledge is a necessary precondition for identifying patients and the periods most

at risk due to the onset of fatigue, so as to be able to hypothesize adequate containment

strategies.

**Setting:** Rizzoli Orthopedic Institute. Department of Chemotherapy

Methods

**Design:** observational study

Population: all patients belonging to the Chemotherapy ward will be recruited

consecutively for a new antiblastic treatment protocol. The process of informing and

collecting the participants' consent will take place during the first admission in which

intravenous administration of the chemotherapy will be started. Potential participants will

be identified / selected for recruitment through inclusion and exclusion criteria described

below. Enrolled patients who will not continue the chemotherapy protocol within our

Institute but at another facility will exit the study.

#### Inclusion criteria:

all patients diagnosed with bone tumors who start a new chemotherapy treatment protocol, both on admission and on an outpatient basis at the Chemotherapy ward for its antiblastic treatment over 12 years of age. The NCCN Guidelines Cancer-Related Fatigue identifies appropriate screening with rating scales with scores from 0 to 10 precisely for patients older than 12 years.

#### **Exclusion criteria:**

patients with little knowledge of the Italian language due to the impossibility of completing the assessment scales.

## **Primary outcome:**

the patient's Fatigue will be measured during the treatment period with antiblastic drugs and part of the followup period. To this end the BFI scale validated in Italian will be used (Mendoza et al 1999; Catania et al, 2013) which includes 9 items with a score for each of 0 to 10 and a consequent total score from 0 to 90. The measurement will take place in 4 times: the day of enrollment, 6 months, 12 months and 24 months after enrollment.

## Secondary outcome:

the quality of life of patients measured by the EORTC QLQ C-30 scale (Aaronson et al, 1993) and the level of autonomy measured by the TESS scale (Davis et al, 1996) in 4 steps: the enrollment day, at 6 months, at 12 months and at 24 months from enrollment.

Variables taken into consideration: through the literature search and the comparison between professionals of different disciplines (nurses, physiotherapists, oncologists) involved, a panel of variables was established to collect:

- Age
- sex
- BMI
- Smoking
- diabetes

- cardiopathies (hypertension, previous heart attack, ...)
- Comorbidity (pulmonary, renal, anemia, arthritis, neuromuscular complications, sleep disorders, pain, emotional distress)
- Diagnosis,
- presence of metastases at the entrance
- type of chemotherapeutic protocol / drug that will be administered from the time of enrollment (Methotrexate, Cisplatin, Adriamycin, Ifosfamide, Elastomer Ifosfamide, Gemcitabine, Taxotere, Vincristine-Adriamycin-ifosfamide, Vincristine phosphamide-Dactomycin, Ifosfamide-etoposide, Temiri, Topotecan, Cyclophosphamide, Eribulin)
- previous chemotherapy treatments: chemotherapy protocol / drugs already performed (Methotrexate, Cisplatin, Adriamycin, Ifosfamide, Elastomer Ifosfamide, Gemcitabine, Taxotere, Vincristine-Adriamycin-ifosfamide, Vincristine phosphamide-Dactomycin, Ifosfamide-etoposide, Temiri, Topotecan, Cyclophosphamide, Eribulina) and number of cycles already carried out.
- number of therapy cycles carried out from the moment of enrollment (to be collected at the 24th month)
- tumor location
- surgery (date and type)
- Perceived pain measured with the NRS scale in the 4 expected data collection times

**Data collection:** the data will be collected at the Chemotherapy ward at the time of admission of the patient in the ward or of his access to the outpatient service. Nurses and the research physiotherapist will be responsible for collecting data by administering the assessment scales and consulting the patient's clinical documentation. Data collection times and specific collection methods are shown in the following tables:

Ver.1.0 del 30/04/2019 5/11

| 1° day | | | |
|------------------------|----------|-----------|-----------|
| DIAGNOSIS/new protocol | | | |
| | | l | |
| Consent/CRF | 6 months | | |
| BFI | BFI | 12 months | |
| QLQ | QLQ | BFI | 24 months |
| TESS | TESS | QLQ | BFI |
| | | TESS | QLQ |
| | | | TESS |

| Variables | Collection methods | Responsible for the collection |
|---|---|---|
| Age | Health documentation - to be included in the enrollment form, then a calculation sheet | Nurse |
| Sex | Health documentation - to be included in the enrollment form, then a calculation sheet | Nurse |
| ВМІ | To be calculated: report the patient's weight and height at the entrance | Nurse |
| Smoking | OBSERVATION sheet (CRF): report in a calculation sheet | Nurse |
| diabetes | OBSERVATION sheet (CRF): report in a calculation sheet | Nurse |
| cardiopathies | OBSERVATION sheet (CRF): report in a calculation sheet | Nurse |
| Diagnosis | Enrollment form: to be reported in the calculation sheet | Nurse |
| presence of | Sanitary documentation: to be included in the | Nurse |

Ver.1.0 del 30/04/2019 6/11

| metastases at the | OBSERVATION (CRF) form, then calculation | |
|---|---|---|
| entrance | sheet | |
| type of | Enrollment form: to be reported in the | Nurse |
| chemotherapeutic | calculation sheet | |
| protocol | | |
| previous | Health documentation - to be included in the | Nurse |
| chemotherapy | enrollment form, then a calculation sheet | |
| treatments | | |
| number of | OBSERVATION sheet (CRF): to be found in | Nurse |
| therapy cycles | health documentation and then in the | |
| | calculation sheet) | |
| tumor location | Enrollment form: to be reported in the | Nurse |
| | calculation sheet | |
| surgery (date and | OBSERVATION sheet (CRF): report in a | Nurse |
| type) | calculation sheet | |
| Pain | Measured with NRS scale. Data present in the | Nurse |
| | BFI Sheet: to be reported in the calculation | |
| | sheet | |
| Autonomy level | TESS scale: self-filled by the patient (6-12-24 | Physiotherapist |
| | months from enrollment) | |

**Statistical analysis**: The characteristics of the sample will be described using the mean and standard or median deviation and interquartile range for quantitative variables and absolute and percentage frequencies for qualitative variables. Simple and multiple linear regression analyzes will be performed and to identify predictors of primary and secondary outcome.

**Sample size:** In a pilot study of 19 patients at the Chemotherapy SSD the average BFI score was 31.6 with DS 19.1 at a mean follow-up of 5.2 months and DS 3.7. On the basis of this data, the number of variables taken into consideration equal to 15 in a multiple linear regression, an effect size of 0.1, an alpha value of 0.05 and a power of 80% the

Ver.1.0 del 30/04/2019 7/11

number of patients to be enrolled is equal to 183. The sample size was calculated with Stata 15.0.

**Duration of the study:** The project lasted 5 years as follows:

Month 1-3 Meeting and training of the team involved in the study

Months 3–36 Patient enrollment and data collection.

Months 36-48 Construction of the database and preliminary analysis

Months 48-60 Follow-up and Statistical analysis of data

The approval date of the Ethics Committee will be considered as the starting date of the trial.

**Safety assessment:** as this is an observational study, patients will be treated in accordance with the rules of good clinical practice and in accordance with the protocols regularly used in the operating unit involved.

Data management and informed consent: the personnel designated by the Investigator must report the information required by the protocol in the CRF form and subsequently in the prepared database. Each potential participant will be fully explained the progress of the study and will be given the opportunity to ask questions and receive answers to all his doubts. The informed consent form must be signed by the participant or a legally authorized representative prior to his participation. Patient documentation must be able to demonstrate that consent was given prior to participation in the study. A copy of the informed consent form must be left to the patient. The consent form, signed by the patient, must be kept at the site.

Approval by the Ethics Committee: This protocol, the informed consent form and all the necessary relevant information related to the study must be submitted to the Ethics Committee for evaluation and must be approved before the start of the study. The study will be conducted in accordance with international standards ISO 14: 155, with the Good Clinical Practice and with the national laws in force.

Ver.1.0 del 30/04/2019 8/11

Confidentiality of data and ownership of results: Adequate documentation will be maintained for everything concerning the patient's clinical data, work sheets, nursing notes; the database will be available in a protected environment and access allowed only with Password. The confidentiality of the patient's sensitive data is guaranteed by the Investigator.

**Publication of Results:** The main investigator undertakes to produce the final report, publish all the data collected as described in the protocol and ensure that the data is reported responsibly and consistently. In particular, the publication of the data deriving from this study will take place regardless of the results obtained. The transmission or diffusion of the data, through scientific publications and / or presentation at congresses, conferences and seminars, will take place exclusively following the merely statistical elaboration of the same, or in any case in an absolutely anonymous form.

# **Bibliografy**

Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76

Araújo JKL, Giglio AD, Munhoz BA, Fonseca FLA, Cruz FM, Giglio AD. Chemotherapy-Induced Fatigue Correlates With Higher Fatigue Scores Before Treatment. Am J Hosp Palliat Care. 2017;34(5):404-411.

Bower JE, Bak K, Berger A, Breitbart W, Escalante CP, Ganz PA, Schnipper HH, Lacchetti C, Ligibel JA, Lyman GH, Ogaily MS, Pirl W F, Jacobsen PB. Screening, assessment, and management of fatigue in adult survivors of cancer: an American Society of Clinical Oncology clinical practice guideline adaptation. J Clin Oncol. 2014 10;32(17):1840-50.

Catania G, Bell C, Ottonelli S, Marchetti M, Bryce J, Grossi A, Costantini M. Cancer-related fatigue in Italian cancer patients: validation of the Italian version of the Brief Fatigue Inventory (BFI). Support Care Cancer. 2013 Feb;21(2):413-9.

Granda-Cameron C, Hanlon AL, Lynch MP, Houldin A. Experience of newly diagnosed patients with sarcoma receiving chemotherapy. Oncol Nurs Forum. 2011 Mar;38(2):160-9. doi: 10.1188/11.ONF.160-169.

Davis AM, Wright JG, Williams JI, et al. (1996) Development of a measure of physical function for patients with bone and soft tissue sarcoma. Qual Life Res, 5:508-16

Hubbard JM, Grothey AF, McWilliams RR, Buckner JC, Sloan JA. Physician perspective on incorporation of oncology patient quality-of-life, fatigue, and pain assessment into clinical practice. J Oncol Pract. 2014 Jul;10(4):248-53.

Mendoza TR, Wang XS, Cleeland CS, et al. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999;85(5):1186–1196.

National Comprehensive Cancer Network (NCCN) Guidelines Version 2.2018

Cancer-related fatigue. https://www.nccn.org/professionals/physician\_gls/pdf/fatigue.pdf.

Accessed 05 Feb 2019

Poort H, Kaal SEJ, Knoop H, Jansen R, Prins JB, Manten-Horst E, Servaes P, Husson O, van der Graaf WTA. Prevalence and impact of severe fatigue in adolescent and young adult cancer patients in comparison with population-based controls. Support Care Cancer. 2017;25(9):2911-2918.

Scott JA, Lasch KE, Barsevick AM, Piault-Louis E. Patients' experiences with cancer-related fatigue: a review and synthesis of qualitative research. Oncol Nurs Forum. 2011 May;38(3):E191-203.

Ver.1.0 del 30/04/2019 10/11

Servaes P, Verhagen S, Schreuder HW, Veth RP, Bleijenberg G. Fatigue after treatment for malignant and benign bone and soft tissue tumors. J Pain Symptom Manage. 2003 Dec;26(6):1113-22.

Stark L, Tofthagen C, Visovsky C, McMillan SC. The Symptom Experience of Patients with Cancer. J Hosp Palliat Nurs. 2012 Jan;14(1):61-70.

Witt J, Murray-Edwards D. Living with fatigue: managing cancer-related fatigue at home and in the workplace. Am J Nurs. 2002 Apr;102 Suppl 4:28-31; quiz 49-52.

Warner JT. Body composition, exercise and energy expenditure in survivors of acute lymphoblastic leukaemia. Pediatr Blood Cancer. 2008 Feb;50(2 Suppl):456-61; discussion 468

Ver.1.0 del 30/04/2019 11/11